CLINICAL TRIAL: NCT03919162
Title: A Phase 2A Randomized Double-Blind Placebo-Controlled Trial to Evaluate the Efficacy and Safety of Varoglutamstat (PQ912) in Patients With Early Alzheimer's Disease With a Stage-Gate to Phase 2B (VIVA-MIND)
Brief Title: A Trial to Evaluate the Efficacy and Safety of PQ912 in Patients With Early AD
Acronym: VIVA-MIND
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: It has been made the strategic decision to terminate the study. This decision to terminate the study early is not being made for safety reasons.
Sponsor: Vivoryon Therapeutics N.V. (Industry)
Collaborators: Alzheimer's Disease Cooperative Study (ADCS) (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PBD-01187; 1R01AG061146-01 (NIH)
Record Dates: First submitted 2019-04-15; First posted 2019-04-18 (Actual); Results first posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's Disease; Mild Cognitive Impairment; Mild Alzheimer's Disease; Early Alzheimer's disease; MCI
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PQ912 (Experimental): All participants started at 150 mg BID and were up-titrated to 600 mg BID
  Interventions: Drug: PQ912
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: PQ912 — PQ912 150 mg tablets
  Other Names: Varoglutamstat
  Arms: PQ912
Other: Placebo — Placebo tablets to mimic PQ912 150 mg tablets
  Arms: Placebo

SUMMARY:
This is a Phase 2A multi-center, randomized, double blind, placebo-controlled, parallel group study of varoglutamstat, with a stage gate to Phase 2B.

In Phase 2A there will be adaptive dosing evaluation of three dose levels with exposure to varoglutamstat or placebo for a minimum of 24 weeks, with preliminary evaluation of both cognitive function and pharmacodynamic changes on EEG spectral analysis in approximately 180 participants.

In the event that the stage gate for Phase 2B is reached, then Phase 2B will assesses efficacy and longer-term safety in a larger study group, i.e., 414.

DETAILED DESCRIPTION:
The goal of this study is to advance a first-in-class, new small molecule treatment for early Alzheimer's disease (AD). Varoglutamstat (PQ912) is an oral, twice daily medication that addresses a novel and significantly differentiated amyloid target: N-terminal post-translationally modified Ab (pGlu-Ab), a particularly toxic subspecies of amyloid beta (Ab).

The study is a Phase 2A multi-center, randomized, double-blind, parallel group trial, with a stage gate to Phase 2B.

This study is conducted to further evaluate whether varoglutamstat's mechanism of action can result in a measurable therapeutic effect on cognition, function and relevant pharmacodynamic (PD) and biological markers in early AD.

Phase 2A is designed to determine the highest dose that is both safe and well tolerated using a predefined Pocock safety stopping boundary based on the rate of adverse events of special interest (AESIs).

During this phase there is an adaptive dosing evaluation with exposure to varoglutamstat or placebo for a minimum of 24 weeks (Phase 2A). Participants are randomized 1:1 to varoglutamstat or placebo, and randomization is stratified between mild AD and MCI, as well as by site.

During Phase 2A participants are to be enrolled sequentially into one of three dose cohorts (labelled Cohort A, B and C, with 60 participants per cohort (n=30 active, n=30 placebo)) and treated at the originally assigned full dose until the Data Safety Monitoring Board (DSMB) provides a protocol-specified dose decision:

Cohort A (600 mg): First 4 weeks 150 mg BID, week 5-8 300 mg BID, week 9-up to 72 600 mg BID;

Cohort B (300 mg): First 4 weeks 150 mg BID, week 5-up to 72 300 mg BID;

Cohort C (150 mg): up to 72 weeks on 150 mg BID.

In addition, at the end of Phase 2A (after 24 weeks) an interim analysis for futility will be conducted evaluating both cognitive function (ADNI Battery Composite score) and pharmacodynamics changes on electroencephalogram (EEG) spectral analysis (EEG theta power) to inform a stage-gate decision on whether to proceed with Phase 2B (72 weeks). If the Phase 2A study meets the predefined criteria to proceed to Phase 2B, then Phase 2B will assess the longer-term efficacy and safety of varoglutamstat in a larger study group, using the dose level determined during Phase 2A. In Phase 2B, a composite cognitive and functional measure as well as PD biomarkers will be used to evaluate efficacy during the extended treatment period.

According to the protocol, during Phase 2A the DSMB performs a continuous review of the safety data using a predefined Pocock safety stopping boundary to provide a dose decision.

If Cohort A does not meet the safety stopping boundary until the last participant of the Cohort A reaches 8 weeks on full dose (600 mg BID) the DSMB will provide a dose decision as per protocol for the dose of Cohort A to be carried forward for all participants in the active arm for the remainder of the study. In case Cohort A meets the stopping boundary, all participants will be down-titrated to the next lower planned dose level (Cohort B) and the same review process by the DSMB will continue until either dose-selection, down-titration to the lowest dose level (Cohort C) or stage-gate decision. As pre-specified, the Pocock safety stopping boundary applies only until dose selection. If the first cohort (Cohort A) with the highest dose of PQ912 (600 mg BID) is selected to be carried forward, evaluation of other dose levels is no longer applicable and all data will be collected as one single active Arm/Group.

All participants randomized to PQ912 will start at 150 mg BID and will be titrated to the dose level selected per protocol; all participants in the placebo group will receive matching placebo. Participants enrolled in Phase 2A remain in the study for seamless inclusion in the Phase 2B evaluation (up to 72 weeks).

ELIGIBILITY:
Key Inclusion Criteria:

* Age 50-89 (inclusive) at screening
* Diagnosed as having Mild Cognitive Impairment (MCI) due to Alzheimer's disease (AD) or Mild probable AD according to workgroups of the Diagnostic Guidelines of the National Institute on Aging and Alzheimer's Association (NIA-AA)
* Mini-Mental State Examination (MMSE) score 20-30 inclusive at screening
* Montreal Cognitive Assessment score (MoCA) < 26 at screening
* Clinical Dementia Rating global score 0.5 or 1 with memory score of > 0.5 at screening
* Positive cerebrospinal fluid (CSF) AD biomarker signature
* A brain MRI scan within 6 months of screening consistent with a diagnosis of Alzheimer's disease
* Participants must have a study partner who has frequent interaction with them (approximately >3-4 times per week), will be present for all clinic visits, and can assist in compliance with study procedures.

Key Exclusion Criteria:

* Significant neurodegenerative diseases and causes of dementia, other than AD, including Parkinson's disease and Huntington's disease, vascular dementia, CJD (Creutzfeldt-Jakob disease), LBD (Lewy Body dementia), PSP (Progressive Supranuclear Palsy), AIDS (Acquired Immunodeficiency Syndrome), or NPH (normal pressure hydrocephalus)
* Meeting Diagnostic Criteria for Possible AD according to workgroups of the Diagnostic Guidelines of the NIA-AA
* Hepatic impairment defined as Child-Pugh class A or more severe liver impairment
* History of moderate or severe skin reactions to medications or current moderate or severe disease of the skin and subcutaneous tissues
* History of a major depressive episode within the past 6 months of screening
* History of diagnosis of schizophrenia
* History of uncontrolled bipolar disorder within past five years of screening
* History of seizures within past two years of screening
* Contraindication to lumbar puncture and MRI
* Monoclonal antibody treatment with anti-amyloid or anti-tau agents intended to address the pathophysiologic processes associated with AD within the previous 180 days prior to baseline (BL)
* Participants who are planning to receive treatment with aducanumab or any Amyloid Beta Antibody during the course of the study
* Participation in another clinical trial for an investigational agent and having taken at least one dose of study drug, unless confirmed as having been on placebo, within 90 days prior to the baseline visit. The end of a previous investigational trial is defined as the date of the last dose of an investigational agent.

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2024-07-12 (Actual); Study Completion 2024-08-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Feldman, Principal Investigator — Alzheimer's Disease Cooperative Study (ADCS)
Locations (22):
- United States (22):
  - Barrow Neurological Institute, Phoenix, Arizona
  - Banner Sun Health Research Institute, Sun City, Arizona
  - The Neuron Clinic, Chula Vista, California
  - University of California, Irvine, California
  - UCSD Alzheimer's Disease Research Center, La Jolla, California
  - Cedars-Sinai Center, Los Angeles, California
  - PCND Neurology, Poway, California
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - USF Health Byrd Alzheimer's Center and Research Institute, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - The University of Iowa Carver College of Medicine, Iowa City, Iowa
  - The University of Kentucky Sanders-Brown Center on Aging, Lexington, Kentucky
  - Northern Light Acadia Hospital, Bangor, Maine
  - NYU Langone Health Tisch Hospital, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Ohio State University, Columbus, Ohio
  - OHSU Neurology Clinic, Portland, Oregon
  - Abington Neurological Associates, Abington, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Lowcountry Center for Veterans Research (LCVR), Charleston, South Carolina
  - UT Health San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Data sharing is integral to the ADCS's (Alzheimer's Disease Cooperative Study) mission to develop and execute innovative clinical trials focused on interventions that may prevent, delay, or treat the expression of Alzheimer's disease and related dementias. The ADCS is committed to sharing resources and tools, including data, biospecimens, trial designs, outcome and analysis measures following NIH guidelines.
  DATA SHARING: The ADCS Data and Sample Sharing Committee (DSSC) grants access to de-identified data to individuals who complete the request process and agree to the conditions in an ADCS/UCSD Data Use Agreement (DUA). After approval and receipt of the fully executed DUA, applicants are authorized to acquire data. Non-compliance with the DUA, including the requirement to provide requested updates will jeopardize further access to data.
Supporting Information: Study Protocol, SAP
Time Frame: January 2026
Access Criteria: Data requestors must complete an ADCS data and sample sharing request form. Upon approval, requestors must complete a data use agreement prior to accessing the data.
URL: https://www.adcs.org/data-sharing/

REFERENCES:
- [Background] Feldman HH, Messer K, Qiu Y, Sabbagh M, Galasko D, Turner RS, Lopez O, Smith A, Durant J, Lupo JL, Revta C, Balasubramanian A, Kuehn-Wache K, Wassmann T, Schell-Mader S, Jacobs DM, Salmon DP, Leger G, DeMarco ML, Weber F; ADCS VIVA-MIND Study Group. Varoglutamstat: Inhibiting Glutaminyl Cyclase as a Novel Target of Therapy in Early Alzheimer's Disease. J Alzheimers Dis. 2024;101(s1):S79-S93. doi: 10.3233/JAD-231126. PMID 39422941
- [Background] Messer K, Jacobs DM, Salmon DP, Qiu Y, Revta C, Weber F, Kuhn-Wache K, Leger GC, Feldman HH. (2022), A novel, efficient and seamless Phase 2A-2B design to test varoglutamstat in early AD: the VIVAMIND study. Alzheimer's Dement., 18(S10): e065197.
- [Background] Lues I, Weber F, Meyer A, Buhring U, Hoffmann T, Kuhn-Wache K, Manhart S, Heiser U, Pokorny R, Chiesa J, Glund K. A phase 1 study to evaluate the safety and pharmacokinetics of PQ912, a glutaminyl cyclase inhibitor, in healthy subjects. Alzheimers Dement (N Y). 2015 Oct 3;1(3):182-195. doi: 10.1016/j.trci.2015.08.002. eCollection 2015 Nov. PMID 29854937
- [Background] Scheltens P, Hallikainen M, Grimmer T, Duning T, Gouw AA, Teunissen CE, Wink AM, Maruff P, Harrison J, van Baal CM, Bruins S, Lues I, Prins ND. Safety, tolerability and efficacy of the glutaminyl cyclase inhibitor PQ912 in Alzheimer's disease: results of a randomized, double-blind, placebo-controlled phase 2a study. Alzheimers Res Ther. 2018 Oct 12;10(1):107. doi: 10.1186/s13195-018-0431-6. PMID 30309389
- [Result] Feldman HH, Messer K, Zhang J, Quach NE, Léger GC, Jacobs DM, Edland SD, Duehring J, MacKelfresh A, Pol A, Revta C, Lupo JL, Balasubramanian A, Lama N, Wassmann T, Schaeffer M, Hoffmann T, Meyer A, Schell-Mader S, Wenzkowski C, Weber F, for the ADCS VIVA-MIND Study Group. The VIVA-MIND study: Topline Results from Phase 2 RCT of Varoglutamstat in Early AD. In press, abstract at 2025 AAIC, Alzheimer's and Dementia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 22 study centers in the US between 2021 and 2024. The first participant was screened on November 10, 2021 and the last participant had his last visit on August 12, 2024. Of 253 screened participants, 112 met inclusion criteria and were randomized to treatment.
Pre-assignment Details: Participants were randomized 1:1 to PQ912 or matching placebo. All participants randomized to PQ912 started at 150 mg BID and were up-titrated to 600 mg BID. Therefore, all data from the participants randomized to PQ912 were collected as one single active Arm/Group and separation of doses is not applicable. Participants enrolled in Phase 2A remained in the study for seamless inclusion in the Phase 2B evaluation (up to 72 weeks). No new participants were enrolled in Phase 2B.
Groups:
- PQ912: All participants started at 150 mg BID and were up-titrated to 600 mg BID administered orally for up to 72 weeks and therefore, all data from these participants were collected as one single active Arm/Group.
  Participants enrolled in Phase 2A remained in the study for seamless inclusion in the Phase 2B evaluation (up to 72 weeks). No new participants were enrolled in Phase 2B.
  PQ912: 150 mg tablets
- Placebo: All participants received matching placebo BID administered orally for up to 72 weeks
  Participants enrolled in Phase 2A remained in the study for seamless inclusion in the Phase 2B evaluation (up to 72 weeks). No new participants were enrolled in Phase 2B.
  Placebo: PQ912 matching placebo tablet
Period: Overall Study
Arm/Group | PQ912 | Placebo
Started | 53 | 59
Treated | 52 | 57
Completed | 13 | 20
Not Completed | 40 | 39
Not completed — Adverse Event | 3 | 2
Not completed — Death | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 12 | 12
Not completed — Study terminated by Sponsor | 20 | 24
Not completed — Screen failure | 1 | 0
Not completed — Missing | 1 | 1

BASELINE CHARACTERISTICS:
Population: The modified intent-to-treat (mITT) population, including all randomized participants who took at least one dose of the study medication and who have a baseline assessment of the primary endpoint for phase 2B (CDR-SB)
Groups:
- Total: Total of all reporting groups
Arm/Group | PQ912 | Placebo | Total
Number analyzed (Participants) | 52 | 57 | 109
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 11 | 19
  >=65 years | 44 | 46 | 90
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72.9 (8.3) | 70.8 (7.4) | 71.8 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 30 | 54
  Male | 28 | 27 | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 50 | 57 | 107
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 4 | 5
  White | 51 | 52 | 103
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 52 | 57 | 109
Alzheimer's Disease Neuroimaging Initiative (ADNI) Battery Composite (ABC) score [Mean (Standard Deviation); unit: Z-scores] — The ABC score was calculated from 9 measures from the ADNI-1 Neuropsychological Test Battery: Auditory Verbal Learning Test (AVLT)-Immediate Recall, AVLT-Delayed Recall, Number Span Forward, Number Span Backward, Category Fluency, Trail Making Test A and, Trail Making Test B, Digit Symbol Substitution, Boston Naming Test. Standardized scores (Z-scores) were calculated using the overall mean and standard deviation of all participants in the mITT at Baseline as reference. The ABC score for each participant was the mean of the standardized subtest values. Range: -3 to 3. Higher scores are better.
  Z-scores | -0.01 (0.65) | 0.00 (0.58) | -0.00 (0.61)
Apolipoprotein E (APOE) genotyping [Count of Participants; unit: Participants] — APOE (E4 +/-) genotype is associated with the risk and age of onset of Alzheimer's disease. Results of APOE genotyping (homozygous or heterozygous for the following alleles: E2, E3, E4) were used to explore a relationship between APOE genotype clinical course and response to treatment. Population: Two patients not included in the denominator for the calculation of percentages because of missing APOE genotype data.
  Participants
    number analyzed (Participants) | 52 | 55 | 107
    E4 carrier - homozygous | 11 | 14 | 25
    E4 carrier - heterozygous | 23 | 30 | 53
    Non-carrier | 18 | 11 | 29
Clinical Dementia Rating - Sum of Boxes (CDR-SB) [Mean (Standard Deviation); unit: Box scores (0-18)] — The CDR-SB scale assesses cognition and daily functioning in patients with Alzheimer's disease across 6 domains (memory, orientation, judgement/problem solving, community affairs, home and hobbies, and personal care). The CDR-SB is a composite rating of cognition and everyday function which incorporates both informant input and direct assessment of performance. Level of impairment in each of the six domains is rated from none (score=0) to severe (score=3). The six domain scores are then summed up to create the CDR-SB. Range: 0-18. Higher scores indicate greater impairment.
  Box scores (0-18) | 3.35 (1.53) | 2.99 (1.70) | 3.16 (1.62)
Quantitative EEG (qEEG) [Mean (Standard Deviation); unit: Proportion (0-1)] — qEEG was used to assess resting-state brain activity, including global relative theta power (4-8 Hz), based on spectral analysis of signals from 21 electrode positions. Higher theta power indicates greater impairment. Population: Only paired EEGs (at least 1 Baseline and 1 Follow-up EEG) were analyzed.
  Proportion (0-1)
    number analyzed (Participants) | 25 | 27 | 52
    (all) | 0.18952 (0.09281) | 0.13596 (0.05351) | 0.16171 (0.07902)
Initial diagnosis [Count of Participants; unit: Participants] — The initial diagnosis of the participant at screening
  Participants
    Mild cognitive impairment due to Alzheimer's disease | 30 | 38 | 68
    Mild probable Alzheimer's disease | 22 | 19 | 41
Site [Count of Participants; unit: Participants] — Sites with 5 or fewer participants included in the mITT population were pooled for analysis
  Participants
    Northern Light Acadia Hospital (AHEMMC) | 5 | 4 | 9
    Banner Sun Health Research Institute (BSHRI) | 4 | 5 | 9
    Northwestern University Feinberg School of Medicine (NWU) | 3 | 5 | 8
    Ohio State University (OSU) | 9 | 8 | 17
    Lowcountry Center for Veterans Research (RJVA) | 3 | 3 | 6
    University of California, Irvine (UCI) | 4 | 3 | 7
    University of California San Diego (UCSD) Alzheimer's Disease Research Center | 4 | 6 | 10
    The University of Iowa Carver College of Medicine (UI) | 5 | 5 | 10
    The University of Kentucky Sanders-Brown Center on Aging (UKY) | 3 | 3 | 6
    Pooled sites | 12 | 15 | 27

OUTCOME MEASURES:

1. Primary Outcome: Phase 2A: Number of Participants With Any Adverse Event of Special Interest (AESI)
Description: The proportion of participants, who experience any AESI during the safety evaluation period, which is from first dose to completion of 8 weeks at the full originally assigned dose. Per protocol, if the first cohort (Cohort A) does not meet the pre-specified Pocock safety stopping boundary within the active arm, that dose will be selected as safe. The dose selected as safe will be the dose carried forward for all participants in the active arm for the remainder of the study. The Pocock boundary is only valid until dose selection. If a higher dose is selected as safe, assignment to lower doses will stop, and all current participants on a lower dose will be titrated up to the selected dose according to uptitration schedule. If Cohort A does not meet the Pocock boundary only evaluation of Cohort A is required for this endpoint.
Time Frame: From first dose to completion of 8 weeks on the full dose (Week 16)
Population: All participants started at 150 mg BID and were up-titrated to 600 mg BID. As pre-specified, this endpoint presents data from first 60 participants (Cohort A) after completion of 8 weeks on full dose, 600 mg BID, because Pocock safety stopping boundary applies only until dose selection.
Measure: Count of Participants; unit: Participants
Groups:
- PQ912: All participants received 600 mg PQ912 BID administered orally for 8 weeks after up-titration period starting with 150 mg BID
- Placebo: All participants received placebo BID administered orally for 16 weeks
Arm/Group | PQ912 | Placebo
Number analyzed (Participants) | 27 | 33
Participants | 1 | 2

2. Primary Outcome: Phase 2A: Median Estimated Target Occupancy (TO) of PQ912 in Cerebrospinal Fluid (CSF) at Week 24
Description: The pharmacokinetics (PK) endpoints in Phase 2A are the derived median values of PQ912 levels in plasma and the corresponding calculated target occupancy (TO) in CSF, following at least 8 weeks of treatment at the dose level being tested. TO in CSF was estimated from plasma PQ912 concentrations.
Time Frame: Week 24, pre-dose (trough level) and 2-3h post-dose
Population: Pharmacokinetic population, including all randomized participants who have received at least 1 dose of the study drug, and who provided sufficient PK samples to reliably estimate 1 plasma PK concentration post-baseline
Measure: Median (Full Range); unit: Percent (%)
Groups:
- PQ912: All participants started at 150 mg BID and were up-titrated to 600 mg BID administered orally for up to 72 weeks and therefore, all data from these participants were collected as one single active Arm/Group
Arm/Group | PQ912
Number analyzed (Participants) | 37
Percent (%)
  Week 24 (Visit 7) - pre-dose | 55.3 [0.0 to 86.4]
  Week 24 (Visit 7) - 2-3h post-dose: number analyzed (Participants) | 24
  Week 24 (Visit 7) - 2-3h post-dose | 94.3 [31.6 to 97.7]

3. Primary Outcome: Phase 2A: Median Plasma Concentrations of PQ912 at Week 24
Description: The pharmacokinetics (PK) endpoints in Phase 2A are the derived median values of PQ912 levels in plasma and the corresponding calculated target occupancy (TO) in CSF, following at least 8 weeks of treatment at the dose level being tested.
  Blood samples were obtained and PQ912 plasma concentrations were determined using a validated high-pressure liquid chromatography hyphenated with tandem mass spectrometry (LC-MS/MS) method.
Time Frame: Week 24, pre-dose (trough level) and 2-3h post-dose
Population: as for outcome 2
Measure: Median (Full Range); unit: ng/mL
Arm/Group | PQ912
Number analyzed (Participants) | 37
ng/mL
  Week 24 (Visit 7) - pre-dose | 208.0 [0.0 to 1070.0]
  Week 24 (Visit 7) - 2-3h post-dose: number analyzed (Participants) | 24
  Week 24 (Visit 7) - 2-3h post-dose | 2790.0 [77.7 to 7210.0]

4. Primary Outcome: Phase 2A: Change From Baseline in Alzheimer's Disease Neuroimaging Initiative (ADNI) Battery Composite (ABC) Score
Description: The within-participant change from baseline in the composite mean of standardized scores from a set of ADNI neuropsychological test measures, the ADNI Battery Composite (ABC, 9-item).
  The ABC score was calculated from the following 9 measures from the ADNI-1 Neuropsychological Test Battery: Auditory Verbal Learning Test (AVLT)-Immediate Recall, AVLT-Delayed Recall, Number Span Forward, Number Span Backward, Category Fluency, Trail Making Test A, Trail Making Test B, Digit Symbol Substitution, Boston Naming Test. Standardized scores (Z-scores) were calculated using the overall mean and standard deviation of all participants in the modified Intent-to-Treat (mITT) population at baseline as reference.
  The ABC score for each participant was the mean of the standardized subtest values. Range: -3 to 3; higher scores indicate less impairment.
Time Frame: 24 weeks
Population: The mITT population, including all randomized participants who took at least one dose of the study medication and who have a baseline assessment of the primary endpoint for phase 2B (CDR-SB)
Measure: Least Squares Mean (Standard Error); unit: Z-scores
Groups:
- Placebo: All participants received matching placebo BID administered orally for up to 72 weeks
Arm/Group | PQ912 | Placebo
Number analyzed (Participants) | 49 | 53
Z-scores | -0.156 (0.036) | -0.214 (0.039)
Statistical Analysis 1: Comparison: PQ912 vs Placebo; Initially after Phase 2A, a futility analysis was planned with a sample size of 90 participants per treatment group to test the 1-sided hypothesis that the rate of decrease of ABC score is greater for the PQ912 group than for the Placebo group. The test should be carried out at a 1-sided 40% significance level, using the mixed effects model. Due to early termination of the study and limited sample size, analysis of Phase 2A data was done in the same manner as final analysis of Phase 2B data; Test type: Superiority; p = 0.2261, Mixed Models Analysis — Null hypothesis was that there was no difference in change of ABC score between the PQ912 and Placebo group after 24 weeks of treatment. P-values <0.05 were considered to be statistically significant; Fixed effect covariates: APOE status, initial diagnosis, site, baseline ABC score, time, treatment group, and time by treatment group interaction; Difference LS Mean = 0.058, 95% CI 2-sided [-0.036 to 0.152], Standard Error of Mean 0.048 — Treatment difference = PQ912 - Placebo

5. Primary Outcome: Phase 2A: Change From Baseline in Quantitative Electroencephalogram (qEEG)
Description: The within-participant change from baseline of global relative theta wave power (4-8 Hz) in qEEG. qEEG was used to assess resting-state brain activity, including global relative theta power (4-8 Hz), based on spectral analysis of signals from 21 electrode positions. Higher theta power indicates greater impairment.
Time Frame: 24 weeks
Population: The modified intent-to-treat (mITT) population, including all randomized participants who took at least one dose of the study medication and who have a baseline assessment of the primary endpoint for phase 2B (CDR-SB). Only paired EEGs (at least 1 evaluable Baseline and 1 evaluable Follow-up EEG) were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Proportion (0-1)
Arm/Group | PQ912 | Placebo
Number analyzed (Participants) | 24 | 25
Proportion (0-1) | 0.01749 (0.00649) | 0.02275 (0.00619)
Statistical Analysis 1: Comparison: PQ912 vs Placebo; Initially after Phase 2A, a futility analysis was planned with a sample size of 90 participants per treatment group to test the hypothesis that increase in EEG theta power is greater for Placebo than for PQ912 (1-sided, alpha = 0.05). Higher theta power is worse; hence this alternative hypothesis indicates benefit of the drug. Due to early termination of the study and limited sample size, analysis of Phase 2A data was done in the same manner as final analysis of Phase 2B data; Test type: Superiority; p = 0.4814, Mixed Models Analysis — Null hypothesis was that there was no difference in change of EEG theta power between the PQ912 and Placebo groups after 24 weeks of treatment. Tests were declared statistically significant if the calculated p-value was ≤ 0.05; Fixed effect covariates: APOE status, initial diagnosis, site, baseline qEEG data, time, treatment group, and time by treatment group interaction; Difference LS Mean = -0.00526, 95% CI 2-sided [-0.02017 to 0.00964], Standard Error of Mean 0.00742 — Treatment difference = PQ912 - Placebo

6. Primary Outcome: Phase 2B: Change From Baseline in Clinical Dementia Rating - Sum of Boxes (CDR-SB) Score
Description: The within-participant change from baseline in CDR-SB scores. The CDR-SB is a composite rating of cognition and everyday function which incorporates both informant input and direct assessment of performance. It assesses through semi-structured interview three cognitive domains (memory, orientation, and judgement/problem solving) and three everyday functional domains (community affairs, home and hobbies, and personal care). Level of impairment in each of the six domains is rated from none (score=0) to severe (score=3). The six domain scores are then summed to create the CDR-SB. Range: 0-18; higher scores indicate greater impairment.
Time Frame: 72 weeks
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: Box scores (0-18)
Groups:
- PQ912: All participants started at 150 mg BID and were up-titrated to 600 mg BID administered orally for up to 72 weeks and therefore, all data from these participants were collected as one single active Arm/Group.
  Participants enrolled in Phase 2A remained in the study for seamless inclusion in the Phase 2B evaluation (up to 72 weeks). No new participants were enrolled in Phase 2B.
- Placebo: All participants received matching placebo BID administered orally for up to 72 weeks.
  Participants enrolled in Phase 2A remained in the study for seamless inclusion in the Phase 2B evaluation (up to 72 weeks). No new participants were enrolled in Phase 2B.
Arm/Group | PQ912 | Placebo
Number analyzed (Participants) | 17 | 22
Box scores (0-18) | 1.63 (0.36) | 1.68 (0.34)
Statistical Analysis 1: Comparison: PQ912 vs Placebo; Null hypothesis is that there was no difference in the change of CDR-SB scores between the PQ912 and the Placebo arms. The primary analysis used a mixed model for repeated measures (MMRM) with within-participant change in CDR-SB score as the outcome. The study planned with 207 participants (including 25% drop-out) per group to have 80% power to detect an effect size of 0.7 points in CDR-SB score. Power calculation was based on a 2-sided t-test with significance level of 0.05; Test type: Superiority; p = 0.9135, Mixed Models Analysis — Tests were declared statistically significant if the calculated p-value is ≤ 0.05; Fixed effect covariates: APOE status, initial diagnosis, site, baseline CDR-SB score, time, treatment group, and time by treatment group interaction; Difference LS Mean = -0.05, 95% CI 2-sided [-1.03 to 0.92], Standard Error of Mean 0.49 — Treatment difference = PQ912 - Placebo

7. Secondary Outcome: Phase 2B: Key Secondary Efficacy: Change From Baseline in Cognitive Functional Composite-2 (CFC2) Score, a Cognitive Functional Composite
Description: The within-participant change from baseline in CFC2 scores. The CFC2 is a novel composite outcome measure of cognition and everyday function that has been derived from measures used in Alzheimer's Disease Neuroimaging Initiative (ADNI) and optimized for detecting change in early Alzheimer's disease (doi.org/10.1016/j.jalz.2012.05.2187). CFC2 is comprised of selected subtests from the Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog) (Word Recall, Delayed Word Recall, and Orientation), Clinical Dementia Rating (CDR) sum of the Cognitive Boxes (Memory, Orientation, Judgement, and Problem Solving), and the Functional Activities Questionnaire (FAQ). The total score for each component subtest was multiplied by -1 so that higher scores indicate better performance. The CFC2 score was then calculated as the sum of the transformed raw scores for the component subtests. Range: -67 to 0; higher scores indicate less impairment.
Time Frame: 72 weeks
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: Total score (-67 to 0)
Arm/Group | PQ912 | Placebo
Number analyzed (Participants) | 16 | 20
Total score (-67 to 0) | -6.694 (1.613) | -7.664 (1.512)
Statistical Analysis 1: Comparison: PQ912 vs Placebo; A hierarchical approach is taken: The key secondary CFC2 follows the primary endpoint (Clinical Dementia Rating - Sum of Boxes), if it is statistically significant, followed by the remaining secondary endpoints in the order defined per Statistical Analysis Plan. Hierarchical testing is stopped as soon as a non-significant result is encountered. If the primary hypothesis is met, then a test for a statistically significant difference will be conducted for the CFC2, however at 4% significance level; Test type: Superiority; p = 0.6528, Mixed Models Analysis — The secondary analysis used a mixed model for repeated measures (MMRM) with the within-participant change compared between active arm and placebo in CFC2 as the outcome; Fixed effect covariates: APOE status, initial diagnosis, site, baseline CFC2, time, treatment group, time by treatment group interaction; Difference LS Mean = 0.969, 95% CI 2-sided [-3.345 to 5.238], Standard Error of Mean 2.140 — Treatment difference = PQ912 - Placebo

8. Secondary Outcome: Phase 2B: Change From Baseline in Alzheimer's Disease Neuroimaging Initiative (ADNI) Battery Composite (ABC, 9-item) Score
Description: The within-participant change from baseline in the composite sum of standardized scores from a set of ADNI neuropsychological test measures, the ADNI Battery Composite (ABC, 9-item). The ABC score is calculated from the following 9 measures from the ADNI-1 Neuropsychological Test Battery: Auditory Verbal Learning Test (AVLT)-Immediate Recall, AVLT-Delayed Recall, Number Span Forward, Number Span Backward, Category Fluency, Trail Making Test A, Trail Making Test B, Digit Symbol Substitution, Boston Naming Test. Standardized scores (Z-scores) were calculated using the overall mean and standard deviation of all participants in the modified intent-to-treat (mITT) population at baseline as reference. The ABC score for each participant was the mean of the standardized subtest values. Range: -3 to 3; higher scores indicate less impairment.
Time Frame: 72 weeks
Population: The modified mITT population, including all randomized participants who took at least one dose of the study medication and who have a baseline assessment of the primary endpoint for phase 2B (CDR-SB)
Measure: Least Squares Mean (Standard Error); unit: Z-scores
Arm/Group | PQ912 | Placebo
Number analyzed (Participants) | 15 | 21
Z-scores | -0.278 (0.078) | -0.378 (0.069)
Statistical Analysis 1: Comparison: PQ912 vs Placebo; A hierarchical approach is taken: If the primary and key secondary endpoint are both statistically significant the remaining secondary endpoints will be tested in the hierarchical order defined per Statistical Analysis Plan until a non-significant result is encountered: Alzheimer's Disease Neuroimaging Initiative (ADNI) Battery Composite Score, Quantitative EEG, Functional Activities Questionnaire, Alzheimer's Disease Assessment Scale - Cognitive Subscale 13, Neuropsychiatric Inventory; Test type: Superiority; p = 0.3241, Mixed Models Analysis — The secondary analysis used a mixed model for repeated measures (MMRM) with the within-participant change compared between active arm and placebo in ABC as the outcome; Fixed effect covariates: APOE status, initial diagnosis, site, baseline ABC score, time, treatment group, time by treatment group interaction; Difference LS Mean = 0.100, 95% CI 2-sided [-0.103 to 0.303], Standard Error of Mean 0.101 — Treatment difference = PQ912 - Placebo

9. Secondary Outcome: Phase 2B: Change From Baseline in Quantitative Electroencephalogram (qEEG)
Description: as for outcome 5
Time Frame: 72 weeks
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Proportion (0-1)
Arm/Group | PQ912 | Placebo
Number analyzed (Participants) | 8 | 10
Proportion (0-1) | -0.01123 (0.01474) | 0.01734 (0.01291)
Statistical Analysis 1: Comparison: PQ912 vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.1398, Mixed Models Analysis — The secondary analysis used a mixed model for repeated measures (MMRM) with the within-participant change compared between active arm and placebo in qEEG as the outcome; Fixed effect covariates: APOE status, initial diagnosis, site, baseline qECG data, time, treatment group, time by treatment group interaction; Difference LS Mean = -0.02857, 95% CI 2-sided [-0.06746 to 0.01032], Standard Error of Mean 0.01846 — Treatment difference = PQ912 - Placebo

10. Secondary Outcome: Phase 2B: Change From Baseline in Functional Activities Questionnaire (FAQ)
Description: The within-participant change from baseline in FAQ.The FAQ is a validated 10-item questionnaire, completed as a structured interview with the study partner, which rates the study participant's ability to carry out ten complex activities of daily living (doi.org/10.1093/geronj/37.3.323). Each item is rated on a scale from 0 (no impairment) to 3 (dependent). Scores are summed across items to provide a total score. Range: 0 to 30; higher scores indicate greater impairment.
Time Frame: 72 weeks
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: Total score (0-30)
Arm/Group | PQ912 | Placebo
Number analyzed (Participants) | 17 | 22
Total score (0-30) | 4.36 (1.35) | 4.97 (1.23)
Statistical Analysis 1: Comparison: PQ912 vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.7377, Mixed Models Analysis — The analysis used a mixed model for repeated measures (MMRM) with the within-participant change compared between active arm and placebo in FAQ as the outcome; Fixed effect covariates: APOE status, initial diagnosis, site, baseline FAQ score, time, treatment group, time by treatment group interaction; Difference LS Mean = -0.60, 95% CI 2-sided [-4.22 to 3.01], Standard Error of Mean 1.79 — Treatment difference = PQ912 - Placebo

11. Secondary Outcome: Phase 2B: Change From Baseline in Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog-13)
Description: The within-participant change from baseline in ADAS-Cog-13. The ADAS-Cog-13 is a structured scale that evaluates memory (immediate and delayed word recall; immediate word recognition), receptive and expressive language, orientation, ideational praxis (preparing a letter for mailing), constructional praxis (copying figures), and attention (number cancellation). Ratings of spoken language, language comprehension, word finding difficulty, and ability to remember test instructions also are obtained. The ADAS-Cog total score is calculated by summing the scores of the 13 component subtests. Range: 0-85; higher scores indicate greater impairment.
Time Frame: 72 weeks
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: Total score (0-85)
Arm/Group | PQ912 | Placebo
Number analyzed (Participants) | 14 | 19
Total score (0-85) | 6.377 (1.627) | 4.343 (1.470)
Statistical Analysis 1: Comparison: PQ912 vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.3496, Mixed Models Analysis — The secondary analysis used a mixed model for repeated measures (MMRM) with the within-participant change compared between active arm and placebo in ADAS-Cog-13 as the outcome; Fixed effect covariates: APOE status, initial diagnosis, site, baseline ADAS-Cog-13 score, time, treatment group, time by treatment group interaction; Difference LS Mean = 2.034, 95% CI 2-sided [-2.292 to 6.360], Standard Error of Mean 2.154 — Treatment difference = PQ912 - Placebo

12. Secondary Outcome: Phase 2B: Change From Baseline in Neuropsychiatric Inventory (NPI)
Description: The within-participant change from baseline in NPI. The NPI is a well-validated, reliable, multi-item instrument to assess psychopathology in Alzheimer's disease dementia based on the results of an interview with the study partner. Frequency and severity of 12 neuropsychiatric symptoms are assessed. Range: 0 to 144; higher scores indicate greater impairment.
Time Frame: 72 weeks
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: Total score (0-144)
Arm/Group | PQ912 | Placebo
Number analyzed (Participants) | 17 | 23
Total score (0-144) | -0.14 (1.80) | 2.95 (1.60)
Statistical Analysis 1: Comparison: PQ912 vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.1933, Mixed Models Analysis — The secondary analysis used a mixed model for repeated measures (MMRM) with the within-participant change compared between active arm and placebo in NPI as the outcome; Difference LS Mean = -3.09, 95% CI 2-sided [-7.81 to 1.62], Standard Error of Mean 2.34 — Treatment difference = PQ912 - Placebo

13. Secondary Outcome: Phase 2B: Assessment of the Longer-term Safety and Tolerability of PQ912 as Measured by Rates of All Treatment-emergent Serious Adverse Events (SAEs)
Description: Longer-term safety and tolerability of PQ912 compared between the active and placebo arm as measured by rates of all treatment-emergent SAEs, presented as numbers of participants with at least one SAE and percentages
Time Frame: 76 weeks
Population: The safety (SAF) population, including all participants who had received at least one dose of the study medication
Measure: Count of Participants; unit: Participants
Groups:
- PQ912: All participants started at 150 mg BID and were up-titrated to 600 mg BID administered orally for up to 72 weeks and therefore, all data from these participants were collected as one single active Arm/Group and separation of doses is not possible.
  Participants enrolled in Phase 2A remained in the study for seamless inclusion in the Phase 2B evaluation (up to 72 weeks). No new participants were enrolled in Phase 2B.
Arm/Group | PQ912 | Placebo
Number analyzed (Participants) | 53 | 56
Participants | 11 | 6

14. Secondary Outcome: Phase 2B: Assessment of the Longer-term Safety and Tolerability of PQ912 as Measured by Suicidality on the Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: Assessment of the longer-term safety and tolerability of PQ912 via the C-SSRS. The C-SSRS is an instrument designed to assess the occurrence, severity, and frequency of suicide-related thoughts and behaviors during the corresponding assessment period. The scale includes suggested questions to elicit the type of information needed to determine if a suicide-related thought or behavior occurred.
  In this study it was used to 'detect' the appearance of new suicidal ideation or behavior as either "present" or "not present". The tables reflect the total number of participants (and percentage) experiencing Any suicidality, Any suicidal ideation, Any suicidal behavior, and Any self-injurious behavior at screening and subsequent time points.
Time Frame: Up to 72 weeks
Population: The safety (SAF) population, including all participants who had received at least one dose of the study medication
Measure: Count of Participants; unit: Participants
Arm/Group | PQ912 | Placebo
Number analyzed (Participants) | 53 | 56
Participants
  Screening - Any suicidality: Present | 3 | 4
  Screening - Any suicidality: Not present | 50 | 52
  Screening - Any suicidal ideation: Present | 3 | 4
  Screening - Any suicidal ideation: Not present | 50 | 52
  Screening - Any suicidal behavior: Present | 1 | 1
  Screening - Any suicidal behavior: Not present | 52 | 55
  Screening - Any self-injurious behavior: Present | 0 | 1
  Screening - Any self-injurious behavior: Not present | 53 | 55
  Baseline - Any suicidality: Present | 4 | 0
  Baseline - Any suicidality: Not present | 49 | 56
  Baseline - Any suicidal ideation: Present | 4 | 0
  Baseline - Any suicidal ideation: Not present | 49 | 56
  Baseline - Any suicidal behavior: Present | 0 | 0
  Baseline - Any suicidal behavior: Not present | 53 | 56
  Baseline - Any self-injurious behavior: Present | 0 | 0
  Baseline - Any self-injurious behavior: Not present | 53 | 56
  Week 4 - Any suicidality: number analyzed (Participants) | 51 | 55
  Week 4 - Any suicidality: Present | 2 | 1
  Week 4 - Any suicidality: Not present | 49 | 54
  Week 4 - Any suicidal ideation: number analyzed (Participants) | 51 | 55
  Week 4 - Any suicidal ideation: Present | 2 | 1
  Week 4 - Any suicidal ideation: Not present | 49 | 54
  Week 4 - Any suicidal behavior: number analyzed (Participants) | 51 | 55
  Week 4 - Any suicidal behavior: Present | 0 | 0
  Week 4 - Any suicidal behavior: Not present | 51 | 55
  Week 4 - Any self-injurious behavior: number analyzed (Participants) | 51 | 55
  Week 4 - Any self-injurious behavior: Present | 0 | 0
  Week 4 - Any self-injurious behavior: Not present | 51 | 55
  Week 8 - Any suicidality: number analyzed (Participants) | 52 | 50
  Week 8 - Any suicidality: Present | 1 | 0
  Week 8 - Any suicidality: Not present | 51 | 50
  Week 8 - Any suicidal ideation: number analyzed (Participants) | 52 | 50
  Week 8 - Any suicidal ideation: Present | 1 | 0
  Week 8 - Any suicidal ideation: Not present | 51 | 50
  Week 8 - Any suicidal behavior: number analyzed (Participants) | 52 | 50
  Week 8 - Any suicidal behavior: Present | 0 | 0
  Week 8 - Any suicidal behavior: Not present | 52 | 50
  Week 8 - Any self-injurious behavior: number analyzed (Participants) | 52 | 50
  Week 8 - Any self-injurious behavior: Present | 0 | 0
  Week 8 - Any self-injurious behavior: Not present | 52 | 50
  Week 12 - Any suicidality: number analyzed (Participants) | 47 | 47
  Week 12 - Any suicidality: Present | 1 | 0
  Week 12 - Any suicidality: Not present | 46 | 47
  Week 12 - Any suicidal ideation: number analyzed (Participants) | 47 | 47
  Week 12 - Any suicidal ideation: Present | 1 | 0
  Week 12 - Any suicidal ideation: Not present | 46 | 47
  Week 12 - Any suicidal behavior: number analyzed (Participants) | 47 | 47
  Week 12 - Any suicidal behavior: Present | 0 | 0
  Week 12 - Any suicidal behavior: Not present | 47 | 47
  Week 12 - Any self-injurious behavior: number analyzed (Participants) | 47 | 47
  Week 12 - Any self-injurious behavior: Present | 0 | 0
  Week 12 - Any self-injurious behavior: Not present | 47 | 47
  Week 16 - Any suicidality: number analyzed (Participants) | 46 | 45
  Week 16 - Any suicidality: Present | 0 | 1
  Week 16 - Any suicidality: Not present | 46 | 44
  Week 16 - Any suicidal ideation: number analyzed (Participants) | 46 | 45
  Week 16 - Any suicidal ideation: Present | 0 | 1
  Week 16 - Any suicidal ideation: Not present | 46 | 44
  Week 16 - Any suicidal behavior: number analyzed (Participants) | 46 | 45
  Week 16 - Any suicidal behavior: Present | 0 | 0
  Week 16 - Any suicidal behavior: Not present | 46 | 45
  Week 16 - Any self-injurious behavior: number analyzed (Participants) | 46 | 45
  Week 16 - Any self-injurious behavior: Present | 0 | 0
  Week 16 - Any self-injurious behavior: Not present | 46 | 45
  Week 24 - Any suicidality: number analyzed (Participants) | 42 | 44
  Week 24 - Any suicidality: Present | 0 | 2
  Week 24 - Any suicidality: Not present | 42 | 42
  Week 24 - Any suicidal ideation: number analyzed (Participants) | 42 | 44
  Week 24 - Any suicidal ideation: Present | 0 | 2
  Week 24 - Any suicidal ideation: Not present | 42 | 42
  Week 24 - Any suicidal behavior: number analyzed (Participants) | 42 | 44
  Week 24 - Any suicidal behavior: Present | 0 | 0
  Week 24 - Any suicidal behavior: Not present | 42 | 44
  Week 24 - Any self-injurious behavior: number analyzed (Participants) | 42 | 44
  Week 24 - Any self-injurious behavior: Present | 0 | 0
  Week 24 - Any self-injurious behavior: Not present | 42 | 44
  Week 36 - Any suicidality: number analyzed (Participants) | 35 | 37
  Week 36 - Any suicidality: Present | 0 | 1
  Week 36 - Any suicidality: Not present | 35 | 36
  Week 36 - Any suicidal ideation: number analyzed (Participants) | 35 | 37
  Week 36 - Any suicidal ideation: Present | 0 | 1
  Week 36 - Any suicidal ideation: Not present | 35 | 36
  Week 36 - Any suicidal behavior: number analyzed (Participants) | 35 | 37
  Week 36 - Any suicidal behavior: Present | 0 | 0
  Week 36 - Any suicidal behavior: Not present | 35 | 37
  Week 36 - Any self-injurious behavior: number analyzed (Participants) | 35 | 37
  Week 36 - Any self-injurious behavior: Present | 0 | 0
  Week 36 - Any self-injurious behavior: Not present | 35 | 37
  Week 48 - Any suicidality: number analyzed (Participants) | 33 | 33
  Week 48 - Any suicidality: Present | 0 | 0
  Week 48 - Any suicidality: Not present | 33 | 33
  Week 48 - Any suicidal ideation: number analyzed (Participants) | 33 | 33
  Week 48 - Any suicidal ideation: Present | 0 | 0
  Week 48 - Any suicidal ideation: Not present | 33 | 33
  Week 48 - Any suicidal behavior: number analyzed (Participants) | 33 | 33
  Week 48 - Any suicidal behavior: Present | 0 | 0
  Week 48 - Any suicidal behavior: Not present | 33 | 33
  Week 48 - Any self-injurious behavior: number analyzed (Participants) | 33 | 33
  Week 48 - Any self-injurious behavior: Present | 0 | 0
  Week 48 - Any self-injurious behavior: Not present | 33 | 33
  Week 60 - Any suicidality: number analyzed (Participants) | 23 | 28
  Week 60 - Any suicidality: Present | 0 | 1
  Week 60 - Any suicidality: Not present | 23 | 27
  Week 60 - Any suicidal ideation: number analyzed (Participants) | 23 | 28
  Week 60 - Any suicidal ideation: Present | 0 | 1
  Week 60 - Any suicidal ideation: Not present | 23 | 27
  Week 60 - Any suicidal behavior: number analyzed (Participants) | 23 | 28
  Week 60 - Any suicidal behavior: Present | 0 | 0
  Week 60 - Any suicidal behavior: Not present | 23 | 28
  Week 60 - Any self-injurious behavior: number analyzed (Participants) | 23 | 28
  Week 60 - Any self-injurious behavior: Present | 0 | 0
  Week 60 - Any self-injurious behavior: Not present | 23 | 28
  Week 72 - Any suicidality: number analyzed (Participants) | 16 | 20
  Week 72 - Any suicidality: Present | 0 | 0
  Week 72 - Any suicidality: Not present | 16 | 20
  Week 72 - Any suicidal ideation: number analyzed (Participants) | 16 | 20
  Week 72 - Any suicidal ideation: Present | 0 | 0
  Week 72 - Any suicidal ideation: Not present | 16 | 20
  Week 72 - Any suicidal behavior: number analyzed (Participants) | 16 | 20
  Week 72 - Any suicidal behavior: Present | 0 | 0
  Week 72 - Any suicidal behavior: Not present | 16 | 20
  Week 72 - Any self-injurious behavior: number analyzed (Participants) | 16 | 20
  Week 72 - Any self-injurious behavior: Present | 0 | 0
  Week 72 - Any self-injurious behavior: Not present | 16 | 20

15. Secondary Outcome: Phase 2B: Assessment of the Longer-term Safety and Tolerability of PQ912 as Measured by Mortality Rates
Description: Longer-term safety and tolerability of PQ912 compared between the active and placebo arm as measured by rates of fatal treatment-emergent serious adverse events (SAEs), presented as numbers of participants with a treatment emergent SAE leading to death and percentages.
Time Frame: 76 weeks
Population: The safety (SAF) population, including all participants who had received at least one dose of the study medication
Measure: Count of Participants; unit: Participants
Arm/Group | PQ912 | Placebo
Number analyzed (Participants) | 53 | 56
Participants | 2 | 0

16. Secondary Outcome: Phase 2B: Assessment of the Longer-term Safety and Tolerability of PQ912 as Measured by Rates of All Treatment-emergent Adverse Events (TEAEs)
Description: Longer-term safety and tolerability of PQ912 compared between the active and placebo arm as measured by rates of all TEAEs, presented as numbers of participants with at least one TEAE and percentages
Time Frame: 76 weeks
Population: The safety (SAF) population, including all participants who had received at least one dose of the study medication
Measure: Count of Participants; unit: Participants
Arm/Group | PQ912 | Placebo
Number analyzed (Participants) | 53 | 56
Participants | 46 | 47

17. Secondary Outcome: Phase 2B: Assessment of the Longer-term Safety and Tolerability of PQ912 as Measured by Rates of All Adverse Events of Special Interest (AESIs)
Description: Longer-term safety and tolerability of PQ912 compared between the active and placebo arm as measured by rates of all AESIs presented as numbers of participants with at least one AESI and percentages .
Time Frame: 76 weeks
Population: The safety (SAF) population, including all participants who had received at least one dose of the study medication
Measure: Count of Participants; unit: Participants
Arm/Group | PQ912 | Placebo
Number analyzed (Participants) | 53 | 56
Participants | 1 | 3

18. Secondary Outcome: Phase 2B: Assessment of the Longer-term Safety and Tolerability of PQ912 as Measured by Drug Discontinuation Rates
Description: Longer-term safety and tolerability of PQ912 compared between the active and placebo arm as measured by rates of drug discontinuation due to treatment-emergent adverse events (TEAEs), presented as numbers of participants with a TEAE leading to drug discontinuation and percentages.
Time Frame: 72 weeks
Population: The safety (SAF) population, including all participants who had received at least one dose of the study medication
Measure: Count of Participants; unit: Participants
Arm/Group | PQ912 | Placebo
Number analyzed (Participants) | 53 | 56
Participants | 6 | 2

ADVERSE EVENTS:
Time Frame: 76 weeks
Description: All participants started at 150 mg BID and were up-titrated to 600 mg BID. As safety data were collected continuously across titration, separation of doses is not possible. Therefore, safety data are reported as one single active Arm/Group. Participants enrolled in Phase 2A remained in the study for seamless inclusion in the Phase 2B evaluation (up to 72 weeks). No new participants were enrolled in Phase 2B.
Groups:
- Placebo: All participants received matching placebo BID administered orally for up to 72 weeks
  Participants enrolled in Phase 2A remained in the study for seamless inclusion in the Phase 2B evaluation (up to 72 weeks). No new participants were enrolled in Phase 2B.
Arm/Group | PQ912 | Placebo
All-Cause Mortality (participants affected / at risk) | 2/53 | 0/56
Serious Adverse Events (participants affected / at risk) | 11/53 | 6/56
Other Adverse Events (participants affected / at risk) | 46/53 | 47/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PQ912 (N=53) | Placebo (N=56)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 1 (2)
Hemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (2)
Bacterial sepsis (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Gastric ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Adverse drug reaction (General disorders) | 0 (0) | 1 (1)
Wound evisceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PQ912 (N=53) | Placebo (N=56)
COVID-19 (Infections and infestations) | 5 (5) | 4 (5)
Nasopharyingitis (Infections and infestations) | 4 (4) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 4 (7)
Diarrhoea (Gastrointestinal disorders) | 9 (9) | 5 (6)
Nausea (Gastrointestinal disorders) | 4 (4) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 8 (12) | 7 (11)
Skin laceration (Injury, poisoning and procedural complications) | 2 (2) | 3 (4)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Depression (Psychiatric disorders) | 1 (1) | 3 (3)
Alanine aminotransferase increased (Investigations) | 1 (1) | 3 (3)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 2 (2) | 4 (5)
Dizziness (Nervous system disorders) | 1 (1) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to the early termination of the study the intended sample size was not reached and the available sample size for the analysis was limited. However, participants enrolled in Phase 2A remained in the study for seamless inclusion in the Phase 2B evaluation (up to 72 weeks).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol (2023-05-17): https://cdn.clinicaltrials.gov/large-docs/62/NCT03919162/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-28): https://cdn.clinicaltrials.gov/large-docs/62/NCT03919162/SAP_001.pdf
  • Informed Consent Form (2023-06-14): https://cdn.clinicaltrials.gov/large-docs/62/NCT03919162/ICF_002.pdf